CLINICAL TRIAL: NCT05595317
Title: The Investigation of the Effects of Non-Immersive Virtual Reality Exercises on Muscle Excitability Around the Knee and Balance in Patients With Knee Osteoarthritis
Brief Title: The Effects of Non-Immersive Virtual Reality Exercises on Muscle Excitability in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Sönmez (Other)
Responsible Party: Sponsor-Investigator, Mehmet Sönmez, Lecturer, Erzurum Technical University
Organization: Erzurum Technical University (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ErzurumTU
Record Dates: First submitted 2022-10-17; First posted 2022-10-26 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis; Virtual Reality
Keywords: Balance; Muscle excitability
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Study group will take Non-immersive Virtual reality (VR) exercise, sham controlled group will take sham VR.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Traditional physiotherapy + A non-immersive virtual reality game will be played to provide treatment for lower limbs.
  Interventions: Device: Non-immersive Virtual Reality
- Sham-controlled group (Sham Comparator): Traditional physiotherapy + A sham non-immersive virtual reality game will be played but not provides treatment for lower limbs.
  Interventions: Device: Sham Non-immersive Virtual Reality

INTERVENTIONS:
Device: Non-immersive Virtual Reality — The traditional physiotherapy program will consist of hot pack (15 minutes), TENS (20 minutes), and 1 set of /10 repetitions of knee flexion/extension exercise for the right and left in a sitting position with hands clasped on opposite shoulders. In the non-immersive virtual reality application, Microsoft Kinect Xbox 360 Adventures games will be applied at the light level exercise level under the supervision of a physiotherapist. The participant will play a game in which he stands in a standing boat in a boat going on a flowing river and has to overcome obstacles by jumping, crouching and stepping left and right (River rush game).
  Other Names: Microsoft Kinect Xbox 360 based therapy; Kinect sensors based therapy; Commercial game consoles based therapy
  Arms: Study group
Device: Sham Non-immersive Virtual Reality — The traditional physiotherapy program will consist of hot pack (15 minutes), TENS (20 minutes), and 1 set of /10 repetitions of knee flexion/extension exercise for the right and left in a sitting position with hands clasped on opposite shoulders. As a sham application, the participants will sit in a chair in front of the screen and try to prevent the balls sent from the opposite direction by using their upper extremities while their bodies are fixed with the help of a belt, under the supervision of a physiotherapist (Rally ball game).
  Other Names: Microsoft Kinect Xbox 360 based sham therapy; Kinect sensors based sham therapy; Commercial game consoles based sham therapy
  Arms: Sham-controlled group

SUMMARY:
The main goal of this sham-controlled clinical trial is to learn the excitability levels of the muscles around the knee and balance using objective measurement methods in patients with knee osteoarthritis of non-immersive virtual reality application. The secondary aims of the study are to investigate in which direction the proprioception, physical function level, independence level in activities of daily living, muscle endurance around the knee and patient satisfaction change with non-immersive virtual reality application in patients with knee osteoarthritis. In this study, main questions are to answer:

1. Are non-immersive virtual reality-based knee exercises effective on muscle excitability around the knee and balance in patients with knee osteoarthritis?
2. Are non-immersive virtual reality-based knee exercises effective in improving the level of physical function in patients with knee osteoarthritis?

The data collection part of this study will be carried out on volunteers, male and female, who have been diagnosed with knee osteoarthritis by a Physical Medicine and Rehabilitation specialist at Erzurum Atatürk University Training and Research Hospital. After informing the participants about the study, the consent form will be signed. Participants will be patients receiving routine outpatient physical therapy. The study was planned as a randomized controlled trial with a sham-control group.

The study group will receive non-immersive virtual reality in addition to traditional physiotherapy, and the control group will receive sham virtual reality exercise in addition to traditional physiotherapy.

DETAILED DESCRIPTION:
Estimated Forty-four volunteer participants with knee osteoarthritis over 18 years who will be at stage of 1-3 according to the Kellgren Lawrence radiological evaluation will be included in the study. The groups will be formed by computerized randomization method after stratification based on gender and knee osteoarthritis severity.

The study group will receive 45 minutes of traditional physiotherapy a day, 5 days a week for 3 weeks, plus 30 minutes of non-immersive virtual reality-based knee joint exercises. The sham-control group will receive 45 minutes of traditional physiotherapy a day, 5 days a week for 3 weeks and 30 minutes of sham non-immersive virtual reality practice.

Demographic data will be evaluated by Demographic Information Form, muscle excitability will be evaluated by superficial Electromyography (EMG) and static balance will be evaluated by Tetrax posturography device. Knee joint proprioception sensation will be achieved with the Protractor and Angle Gauge (Toolkit, Korea) application. Physical function assessment with Western Ontario and McMaster Universities Arthritis Index (WOMAC), independence level with Katz Activities of Daily Living Independence Index, muscular endurance with 30-second stand-up test (30 Seconds Chair Stand Test), dynamic balance with Timed Up and Go test, Participants' satisfaction with the treatment they receive will be evaluated with a 10-centimeter Visual Analogue Scale (VAS). Measurements will be performed at baseline and at the end of the 3rd week of treatment as post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Those over the age of 18
* Those with a Kellgren and Lawrence score between 1-3
* Those who can walk > 15 m independently
* Those who agreed to participate in the study.

Exclusion Criteria:

* Those with knee osteoarthritis with any contagious infection, autoimmune disease or fracture
* Those with a history of malignancy, dizziness, vertigo or stroke that may affect posture and balance, or a history of underlying neurological and vestibular disease
* Those who have undergone any knee operation
* Those receiving injection therapy for knee OA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-10-29 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
Muscle Excitability | Change from baseline muscle excitability at week 3.
  Electromyography will be used to evaluate muscle excitability. Superficial electrodes will be used for assessments, no needle electrodes will be used.
  EMG or ENMG (electroneuromyography); It is expressed by the abbreviation of the terms electro (electrical), neuro (nerve), myo (muscle) and graphy (writing). Electromyography is a test used to measure the natural electrical activity of muscles. It can be determined that the disease, which is evaluated by EMG, originates from the muscle or nervous system. During the EMG process, the signals coming from the muscles and nerves are transferred to the digital environment as data through a special device and electrodes. The data in the digital environment are interpreted by neurologists and it is evaluated whether there is any abnormality. EMG is divided into two applications: surface EMG, where the electrodes are attached to the skin, and needle EMG, where the needle electrode is inserted into the muscle.
Static Balance | Change from baseline static balance at week 3.
  The Tetrax® Interactive Static Posturography System (Tetrax°) (Sunlight Medical Ltd, Israel) will be used to assess static balance.
  It is a computerized posturography measuring device that is frequently used in the measurement of static balance. A total of 8 different measurements are made, with eyes open and closed. Eight different postures are evaluated for the test, and each posture is measured for 32 seconds. Initial stance, head up, eyes open (NO), then head upright, eyes closed (NC) stance is evaluated to limit visual impact; thereby emphasizing the influence of the somatic sense or vestibular organ. Next, four different postures are tested in the following order: head to the right (HR), head turned 45° to the right; head left (HL), head turned 45° left; Measurements are completed with the head back (HB), tilting the head back 30° and facing the ceiling, and forward (HF), tilting the head forward 30° and facing the floor.

SECONDARY OUTCOMES:
Knee Proprioception | Change from baseline knee proprioception at week 3.
  Protractor and Angle Gauge (Toolkit, Korea) will be used to evaluate knee proprioception.It is a free phone application that evaluates by measuring the angular changes precisely by marking the joints through an application.
Physical Function Level | Change from baseline Physical Function Level at week 3.
  Physical function level will be assessed with Western Ontario and McMaster Universities Arthritis Index (WOMAC) Turkish version. It is a scale that evaluates the disability associated with these conditions in hip and/or knee osteoarthritis. It consists of three parts: pain, stiffness and physical function. It contains a total of 24 items. Items are scored on a Likert scale. The degree of pain and strain is indicated by giving points from 0 to 4 on the Likert scale. Total score can be between 0-96 points. Higher score indicates worse functional level.
Independence in Activities of Daily Living | Change from baseline Independence in Activities of Daily Living at week 3.
  KATZ Index Turkish version will be used to evaluate Independence in Activities of Daily Living. It determines the independence levels of the participants in 6 different areas: bathing, dressing, toileting, transfer, continence and feeding. It is scored from 0 to 6 points. 0 means dependent, 6 means fully independent.
Muscle Endurance | Change from baseline Endurance at week 3.
  The muscle endurance will be measured with 30 Seconds Chair Stand Test. It is a test that evaluates the participant's sitting and standing endurance. The number of sit-ups performed during 30 seconds is recorded. If it is less than 10, the endurance is considered insufficient.
Dynamic Balance | Change from baseline Dynamic Balance at week 3.
  Dynamic balance measurement will be performed by using Timed Up and Go test.This test requires a standard chair, a stopwatch, and a 3-metre hole. The participant gets up from the chair at the command and returns from the marked point 3 meters ahead, sits on the chair and the time is recorded. If it is longer than 12 seconds, it is said that there is a dynamic balance disorder.
Patient Satisfaction from Treatment | At week 3.
  Visual Analogue Scale will be used to evaluate patient satisfaction regarding treatment. This scale is found by measuring the distance of the marked point with the help of a ruler after the participant randomly marks any point on a 10 cm long horizontal line. On the line, the leftmost point is marked as dissatisfied, and the rightmost point is marked as very satisfied with the treatment. Participants mark any point above or between these two points. Higher score show more satisfaction level.

CONTACTS AND LOCATIONS:
Overall Officials: Şebnem AVCI, PhD, Study Director — Abant Izzet Baysal University
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No